CLINICAL TRIAL: NCT02939495
Title: The Efficacy and Safety of Dapoxetine/Sildenafil Combination Therapy in the Treatment of Men With Premature Ejaculation and Erectile Dysfunction (DAP-SPEED Study)
Brief Title: The Efficacy and Safety of Dapoxetine/Sildenafil Combination Therapy
Acronym: DAP-SPEED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Neutec Ar-Ge San ve Tic A.Ş (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEU-16.12; 16-NEU-1 (Other: Ministry of Health, Turkey)
Record Dates: First submitted 2016-08-20; First posted 2016-10-20 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Premature Ejaculation; Erectile Dysfunction
Keywords: Premature Ejaculation; Erectile Dysfunction; DAP-SPEED; Dapoxetine; Sildenafil
MeSH Terms: conditions — Premature Ejaculation; Erectile Dysfunction | interventions — dapoxetine; Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study drug (Experimental): Dapoxetine/Sildenafil 30/50 mg film coated tablet
  Interventions: Drug: Dapoxetine/Sildenafil 30/50 mg film coated tablet

INTERVENTIONS:
Drug: Dapoxetine/Sildenafil 30/50 mg film coated tablet — 1 tablet before sexual intercourse
  Other Names: Dapoxil

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Dapoxetine/Sildenafil 30/50 mg film-coated tablet in the treatment of men with premature ejaculation and erectile dysfunction.

DETAILED DESCRIPTION:
During 4-weeks treatment period, patients will take one Dapoxetine/Sildenafil 30/50 mg film coated tablet 1-3 hours before sexual intercourse.

Study drug should not be used more than 1 tablet every 24 hours during the treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years old men,
* Participants must be heterosexual males and in a stable monogamous sexual relationship with a female partner for at least 6 months and will continue throughout the study,
* Clinical diagnosis of erectile dysfunction, IIEF score ≤21,
* Premature Ejaculation Diagnostic Tool (PEDT) score must be ≥11
* Patients with life-long PE and acquired PE according to the description of International Society for Sexual Medicine (ISSM) ,
* The patient and his partner must have sexual intercourse twice a week for the duration of the study,
* Commitment to comply with the study protocol,
* Patients who sign informed consent form (ICF).

Exclusion Criteria:

* History of medical events such as surgical interventions or neurologic conditions (e.g., multiple sclerosis), trauma, or infections that are associated with the development of symptoms of premature ejaculation (PE) and considered a potential cause of PE,
* Having genital abnormalities, except penile curvature unless not prevent sexual intercourse,
* Developed ED or PE due to drug use or quit taking drugs,
* Any conditions that prevent sexual intercourse with partners
* History of epilepsy,
* Severe renal insufficiency,
* Liver disease,
* History of in last 6 months stroke, myocard infarction, cardiac insufficiency (New York Cardiovascular Associates (NYCA) phase II-IV), AV block or message disorder such as sick sinus syndrome, severe ischemic cardiac disease, syncope, unstable angına, life-threatening arrhythmia or hypotension,
* Non-Arteritic Anterior ischemic optic neuropathy,
* Patients who are not eligible to have sexual intercourse due to existing health problems,
* Autonomic neuropathy, retinitis pigmentosa, blood diseases, active peptic ulcer, abnormalities in ECG, severe systemic disease that cannot be controlled,
* Systolic/Diastolic blood pressure at rest <90/50mmHg and 170/100mmHg<
* History of allergy to Selective Serotonine Reuptake Inhibitor (SSRI) and phosphodiesterase inhibitor drugs,
* Continuing to use or quitted in last 3 months of Monoamine oxidase inhibitor (MAOI), Thioridazine, Serotonine Reuptake Inhibitor (SSRI), Selective-Norepinephrin Reuptake Inhibitor (SNRI), Serotonergic drug/herbal product, tricyclic antidepressant and atypical antipsychotic drugs,
* Use of nitrates, alfa blockers, vasodilators, ketoconazole, itraconazole, ritonavir, saquinavir, telithromycin, nefazodone, nelfinavir, atazanavir, cimetidine, erithromicin, clarithromycin, fluconazole, amprenavir, fosamprenavir, aprepitant, verapamil, diltiazem, any kind of vasodilator, antiplatelet, anticoagulant, dapoxetine, PDE5 inhibitor, alcohol and stimulant drug,
* Patients on a different therapy (behavioral therapy or other drugs that are applied locally) for PE treatment
* During the study, the possibility of taking medication which may affect the study drug's pharmacokinetic/pharmacodynamic properties
* Patients who are defining symptoms of prostatitis clinically
* Thyroid hormone disorders

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
The evaluation of change in Intra-vaginal Ejaculation Latency Time (IELT) compared to baseline. | 4-weeks
The evaluation of IIEF-15 (International Index of Erectile Function Questionnaire) score compared to baseline. | 4-weeks
The evaluation of premature ejaculation symptom scores compared to baseline. | 4-weeks

SECONDARY OUTCOMES:
The evaluation of Premature Ejaculation response measured by Premature Ejaculation Profile (PEP) | 4-weeks
The Rate of Premature Ejaculation Profile (PEP) response | 4-weeks
The evaluation of safety of study drug (Number of Participants with Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment) | 4-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ege Can Şerefoğlu, Assoc Prof Dr, Principal Investigator — Bahçeci Grup
Locations (1):
- Bagcilar Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Tuken M, Culha MG, Serefoglu EC. Efficacy and safety of dapoxetine/sildenafil combination tablets in the treatment of men with premature ejaculation and concomitant erectile dysfunction-DAP-SPEED Study. Int J Impot Res. 2019 Mar;31(2):92-96. doi: 10.1038/s41443-019-0122-2. Epub 2019 Jan 31. PMID 30705437